CLINICAL TRIAL: NCT07271186
Title: A Phase 2 Randomized, Double-Blind, Placebo-Controlled Study to Assess the Efficacy, Safety, Pharmacokinetics, and Pharmacodynamic Effects of ANGPTL3 Inhibition With Either Small-Interfering RNA Alone or in Combination With an ANGPTL3 Antibody in Participants With Diabetic Kidney Disease
Brief Title: Study to Assess the Effects of Angiopoietin-like Protein 3 (ANGPTL3) Inhibition in Adult Participants With Diabetic Kidney Disease
Acronym: ANCHOR-POC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALN-ANG3-CKD-2502
Record Dates: First submitted 2025-11-21; First posted 2025-12-09 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Diabetic Kidney Disease (DKD)
Keywords: Chronic Kidney Disease (CKD); Type 2 Diabetes; Lipid Management
MeSH Terms: conditions — Diabetic Nephropathies; Renal Insufficiency, Chronic; Diabetes Mellitus, Type 2 | interventions — evinacumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- ALN-ANG3 + evinacumab placebo (Experimental)
  Interventions: Drug: ALN-ANG3; Drug: Evinacumab placebo
- ALN-ANG3 + evinacumab (Experimental)
  Interventions: Drug: ALN-ANG3; Drug: Evinacumab
- ALN-ANG3 placebo + evinacumab placebo (Placebo Comparator)
  Interventions: Drug: ALN-ANG3 placebo; Drug: Evinacumab placebo

INTERVENTIONS:
Drug: ALN-ANG3 — Administered per the protocol
  Arms: ALN-ANG3 + evinacumab; ALN-ANG3 + evinacumab placebo
Drug: Evinacumab — Administered per the protocol
  Other Names: Evkeeza®; R1500
  Arms: ALN-ANG3 + evinacumab
Drug: ALN-ANG3 placebo — Administered per the protocol
  Arms: ALN-ANG3 placebo + evinacumab placebo
Drug: Evinacumab placebo — Administered per the protocol
  Arms: ALN-ANG3 + evinacumab placebo; ALN-ANG3 placebo + evinacumab placebo

SUMMARY:
This study is researching experimental drugs called ALN-ANG3 and evinacumab (called "study drugs"). The study is focused on participants who have diabetic kidney disease.

The aim of the study is to see how safe and effective the study drugs are.

The study is looking at several other research questions, including:

* What side effects may happen from taking the study drug
* How much study drug is in the blood at different times

ELIGIBILITY:
Key Inclusion Criteria:

1. Medical history of type 2 diabetes and receiving medical therapy or lifestyle interventions for glucose management
2. Hemoglobin A1C (HbA1c) of 6.5 to 10% at screening
3. eGFR 30 to 90 mL/min/1.73 m^2 using 2021 Chronic Kidney Disease-Epidemiology Collaboration-Estimated Glomerular Filtration Rate using Creatinine and Cystatin C (CKD-EPI eGFRcr-cys) equation at screening
4. Albuminuria: Urine Albumin to Creatinine Ratio (UACR) of 500 to 5000 mg/g at screening

Key Exclusion Criteria:

1. Known medical history or clinical evidence indicative of non-diabetic renal disease
2. Renal disease that required treatment with systemic immunosuppressive therapy, or a history of dialysis or renal transplant
3. Medically unstable as assessed by the investigator
4. Hospitalization (ie, >24 hours) within 30 days of the screening visit

NOTE: Other Protocol-Defined Inclusion/Exclusion Criteria Apply

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2026-01-09 (Actual); Primary Completion 2027-09-24 (Estimated); Study Completion 2028-04-07 (Estimated)

PRIMARY OUTCOMES:
Percent change in Urine Albumin to Creatinine Ratio (UACR) | Baseline to Week 24

SECONDARY OUTCOMES:
Change in Estimated Glomerular Filtration Rate (eGFR) | Baseline to Week 24
Change in total cholesterol | Baseline to Week 24
Change in Low-Density Lipoprotein-Cholesterol (LDL-C) | Baseline to Week 24
Change in High-Density Lipoprotein-Cholesterol (HDL-C) | Baseline to Week 24
Change in non-High-Density Lipoprotein-Cholesterol (non-HDL-C) | Baseline to Week 24
Change in triglycerides | Baseline to Week 24
Change in Apolipoprotein B (ApoB) | Baseline to Week 24
Concentration of combined ALN-ANG3 and metabolite(s) and evinacumab | Up to Week 24
Change in concentration of Angiopoietin-Like Protein-3 (ANGPTL-3) | Baseline to Week 24
Occurrence of Treatment-Emergent Adverse Events (TEAEs) | Up to Week 48
Severity of TEAEs | Up to Week 48
Incidence of ADAs to ALN-ANG3 | Through Week 24
Magnitude of ADAs to ALN-ANG3 | Through Week 24
Incidence of ADAs to evinacumab | Through Week 24
Magnitude of ADAs to evinacumab | Through Week 24

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (10):
- United States (10):
  - Applied Research Center of Arkansas, Little Rock, Arkansas
  - Amicis Research Center, Northridge, California
  - Amicis Research Center, Santa Clarita, California
  - Amicis Research Center, Valencia, California
  - Elixia Hollywood, Hollywood, Florida
  - Research by Design, LLC - Internal Medicine, Chicago, Illinois
  - Elixia MNA, City of Saint Peters, Missouri
  - Clinical Research Consultants, LLC, Kansas City, Missouri
  - Northeast Clinical Research Center, Bethlehem, Pennsylvania
  - Suburban Research Associates, West Chester, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has:
  * received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication or has globally discontinued development of the product for all indications on or after April 2020 and has no plans for future development
  * made the study results publicly available (e.g., scientific publication, scientific conference, clinical trial registry)
  * the legal authority to share the data, and
  * ensured the ability to protect participant privacy
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/